CLINICAL TRIAL: NCT03557541
Title: Sardine-enriched Diet for Prevention Type 2 Diabetes in Elderly and Prediabetic Population
Brief Title: Sardine-enriched Diet for Prevention Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Principal Investigator, Diana Alicia Diaz Rizzolo, RD, Msc, PhD candidate, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/8863
Record Dates: First submitted 2018-03-21; First posted 2018-06-15 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes; Diet Habit; Diabetes; Nutritional and Metabolic Disease
Keywords: diabetes; T2D; diet; nutrition; prediabetes; sardine; elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Feeding Behavior; Diabetes Mellitus; Metabolic Diseases | interventions — calcitonin, sardine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sardine group (Experimental)
  Interventions: Dietary Supplement: Sardine
- Control group (Active Comparator)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Sardine — They received 200gr of canned sardine in olive oil per week (+a common T2D-preventive diet)
  Arms: Sardine group
Dietary Supplement: Control — They received a common T2D-preventive diet
  Arms: Control group

SUMMARY:
The hypothesis formulated is that 200 g of sardine on a weekly basis will have a favourable impact avoiding the natural development of the pathology due to changes in the biochemical profile, the anthropometrics, inflammatory markers, changes in gut microbiota populations, also in transcriptomics and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* glycaemia between 100-125 md / dL or ≥5.7% HbA1c

Exclusion Criteria:

* treatment with oral antidiabetic drugs
* any nutritional education to prevent T2D
* Suspect or known hypersensitivity to sardine or related fish
* Chronic treatment with oral steroids and / or AINES
* Treatment with oral antidiabetic agents and / or insulin
* Treatment with immunosuppressive drugs
* Diagnosis of active neoplasm
* Diagnosis of HIV or AIDS
* Abnormal liver profile (> 6 times normal values)
* Diagnosis of Acute Psychiatric Sdr
* Presence of serious acute concomitant disease, which it requires more than 7 days of recovery.
* Major cardiovascular event (stroke, myocardial infarction) in the month prior to randomization.
* Any other condition that the investigator considers to be inoperative so that the subject conducts the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
type 2 diabetes new onset | Change from Baseline at 12 months
  incidence of new diagnosis of type 2 diabetes

SECONDARY OUTCOMES:
adiponectin | Change from Baseline at 12 months
  adiponectin levels
quantification of gut microbiota populations | Change from Baseline at 12 months
  quantification by q-PCR
gene expression | Change from Baseline at 12 months
  relative expression related genes by RT q-PCR (Real Time Quantitative Reverse transcription polymerase chain reaction)
metabolomics study of dietary biomarkers and health biomarkers [(1) Fatty acyls, bile acids, steroids and lysoglycerophospholipids, (2) Glycerolipids, glycerophospholipids, sterol lipids and sphingolipids, (3) Amino acids.] | Change from Baseline at 12 months
  endogenous metabolic profiles of serum samples will be studied using ultra-high performance liquid chromatography - mass spectrometry (UHPLC-MS). The same unit for measurements [log2 (fold change)]
glucose homeostasis | Change from Baseline at 12 months
  glucose (mg/dl)
insulin levels | Change from Baseline at 12 months
  insulin (mU/L)
HOMA-IR (homeostasis model assessment insulin resistance) | Change from Baseline at 12 months
  insulin resistance index
HOMA-B (homeostasis model assessment B cell function) | Change from Baseline at 12 months
  B cella function

CONTACTS AND LOCATIONS:
Locations (1):
- Diana A Diaz Rizzolo, Barcelona, Spain

REFERENCES:
- [Derived] Diaz-Rizzolo DA, Serra A, Colungo C, Sala-Vila A, Siso-Almirall A, Gomis R. Type 2 diabetes preventive effects with a 12-months sardine-enriched diet in elderly population with prediabetes: An interventional, randomized and controlled trial. Clin Nutr. 2021 May;40(5):2587-2598. doi: 10.1016/j.clnu.2021.03.014. Epub 2021 Mar 18. PMID 33932804

DOCUMENTS (2):
  • Informed Consent Form (2013-11-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03557541/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2013-11-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03557541/Prot_SAP_001.pdf